CLINICAL TRIAL: NCT00871507
Title: SD in Subjects With T2DM
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics (Explores What the Body Does to the Drug), and Pharmacodynamics (Explores What a Drug Does to the Body) of JNJ-38431055 in Volunteers With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR016048
Record Dates: First submitted 2009-03-26; First posted 2009-03-30 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 001 (Experimental)
  Interventions: Drug: JNJ-38431055 Dose 1
- 002 (Experimental)
  Interventions: Drug: JNJ-38431055 Dose 2
- 003 (Placebo Comparator)
  Interventions: Drug: Placebo
- 004 (Active Comparator)
  Interventions: Drug: Sitagliptin 100 mg

INTERVENTIONS:
Drug: JNJ-38431055 Dose 1 — Liquid suspension/solution of JNJ-38431055 administered as a single dose
  Arms: 001
Drug: Sitagliptin 100 mg — Capsule containing 100 mg of sitagliptin administered as a single dose.
  Arms: 004
Drug: Placebo — Placebo suspension/solution and Placebo capsule administered as single doses
  Arms: 003
Drug: JNJ-38431055 Dose 2 — Liquid suspension/solution of JNJ-38431055 administered as a single dose
  Arms: 002

SUMMARY:
This study will assess the safety, tolerability, pharmacokinetics (explores what the body does to the drug), and pharmacodynamics (explores what a drug does to the body) of JNJ-38431055 in volunteers with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
This is a double-blind (neither physician or participant knows name of the assigned study drug), placebo-controlled (substance containing no medication), crossover study in male and female volunteers with type 2 diabetes mellitus. For each volunteer, the study consists of a screening phase (up to 45 days), a run-in phase during which volunteers discontinue their oral hypoglycemic drugs (28 days), a treatment phase during which volunteers will continue to be off their oral hypoglycemic drugs (28 days) and will receive 4 single dose study treatments in a randomized (study sequence assigned by chance) sequence, and a follow-up phase (10 days). After the follow-up phase volunteers will restart their oral hypoglycemic drugs. During the treatment phase there will be at least 7 days between each of the 4 treatments. The four treatments will be Dose 1 of JNJ-38431055, Dose 2 of JNJ-38431055, sitagliptin (Januvia), and placebo. The following safety evaluations will be taken throughout the study: Electrocardiogram (an ECG is a painless procedure that gives a picture of the electrical activity of the heart), Blood pressure, heart rate, and blood samples for laboratory tests. The primary outcome will be incremental glucose after an oral glucose tolerance test. Study drug will be administered as single oral doses separated by at least 7 days. The four treatments will be Dose 1 of JNJ-38431055, Dose 2 of JNJ-38431055, sitagliptin (Januvia), and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Males or postmenopausal or surgically sterilized females, who have type 2 diabetes mellitus
* Medically stable on the basis of physical examination, medical history, laboratory safety test results, vital signs and ECG performed at Screening
* Body Mass Index (BMI) between 22 and 39.9 kg/m2, inclusive
* On a generally stable antihyperglycemic agent regimen (i.e., with no change in medication, or only 1 dose step change in dose) for at least 2 months prior to the Screening Visit, including volunteers who are:(a) Not currently on antihyperglycemic therapy and have an HbA1c =7.0% and =10.0%, or (b) On a single oral antihyperglycemic agent [metformin, a sulfonylurea, a meglitinide (e.g., repaglininide or nateglinide), a DPP-4 inhibitor (sitagliptin or vildagliptin), or an alpha-glucosidase inhibitor (e.g., acarbose)] and have an HbA1c >=6.5% and <=9.5%, or (c) On low-dose dual oral agent therapy (i.e., <50% maximum labeled doses of both agents) and have an HbA1c >=6.5% and <=9.5%
* On Day -1, FPG concentrations between 120 mg/dL and 260 mg/dL, inclusive.

Exclusion Criteria:

* Taking non-oral antihyperglycemic agent (e.g., insulin, exenatide or other GLP-1 analogues), or taking a thiazolidinedione (i.e., a PPARg agonist) within 3 months of Day -1
* History of a recent severe hypoglycemic episode, recurrent hypoglycemic episodes (i.e., within the past year), or a history of hypoglycemic unawareness
* History of clinically significant diabetic complications, including retinopathy, nephropathy, neuropathy or gastroparesis
* Positive test for alcohol and/or drugs of abuse
* Psychological and/or emotional problems, which would render the informed consent invalid, or limit the ability of the volunteer to comply with the study requirements
* Any condition that, in the opinion of the investigator, would compromise the well being of the volunteer or the study or prevent the volunteer from meeting or performing study requirements.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2009-04; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Incremental glucose AUC after an oral glucose tolerance test (OGTT) | 0-4 hours after OGTT

SECONDARY OUTCOMES:
Incremental glucose AUC after a meal tolerance test (MTT) | 0-4 hours after MTT
Measurements of beta-cell function | 0-4 hours after OGTT/MTT
Effect on incretin levels | 0-4 hours after OGTT
Pharmacokinetics | 48 hours after dosing
Safety and Tolerability | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (2):
- United States (2):
  - Fort Myers, Florida
  - San Antonio, Texas